CLINICAL TRIAL: NCT02704130
Title: Transarterial Embolization and Microwave Ablation Combination Therapy in Early-stage Hepatocellular Carcinoma: A Randomized Trial
Brief Title: TAE and MWA Combination Therapy in Early-stage Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-16-23B
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Liver Cancer, Adult; Liver Cell Carcinoma; Liver Cell Carcinoma, Adult
Keywords: Therapeutic Embolization; Ablation Techniques; Transarterial Embolization; TAE; Microwave Ablation; MWA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TAE + MWA combination therapy (Experimental): In patients randomized to receive the experimental therapy, transarterial embolization (TAE) treatments will be initiated within one week of randomization. Blunt embolization will be performed with LC beads with a maximum size of 700 µm. Microwave ablation (MWA) will be performed up to one month following randomization. The LC beads will be admixed with 8-15 mL of contrast and injected into the arterial branch at a rate of 1-2 mL/min. Treatment may be discontinued if any exclusion criteria develop in the patient or at the patient's request.
  Interventions: Device: Transarterial embolization; Procedure: Microwave Ablation
- MWA monotherapy (Active Comparator): Microwave ablation (MWA) will be performed up to one month following randomization. Treatment may be discontinued if any exclusion criteria develop in the patient or at the patient's request. All operative MWAs will be performed in a laparoscopic or robot-assisted laparoscopic setting. All ablations will be guided by intraoperative ultrasound. Ablations will be performed with a 2.45-GHz generator with a 1.8-mm-diameter transcutaneous antenna.
  Interventions: Procedure: Microwave Ablation

INTERVENTIONS:
Device: Transarterial embolization — In transarterial bland embolization, beads are delivered directly into the arterial vessels feeding the tumor, usually by a percutaneous coaxial catheter system guided by ultrasound or fluoroscopy through the common femoral artery.
  Other Names: TAE
  Arms: TAE + MWA combination therapy
Procedure: Microwave Ablation — Microwave ablation is a form of thermal ablation used to treat cancer. In this procedure, electromagnetic waves in the microwave energy spectrum (300 MHz to 300 GHz) are applied to tumor tissue. The oscillation of polar molecules produces frictional heating, ultimately generating tissue necrosis within solid tumors.

SUMMARY:
This is a single-center, prospective RCT to study the effectiveness of TACE and MWA combination therapy with MWA monotherapy for the treatment of early HCC. Primary outcome is 2-year intrahepatic disease-free survival.

DETAILED DESCRIPTION:
This single-center, prospective randomized controlled trial (RCT) is designed to compare the outcomes and clinicopathologic results of trans arterial embolization (TAE) and microwave ablation (MWA) combination therapy with MWA monotherapy for the treatment of early (stages 0 and A) hepatocellular carcinoma (HCC). The primary aim of this study is to test the following hypothesis: 2-year intrahepatic disease-free survival does not differ between patients receiving the experimental therapy (MWA + TAE) and patients receiving the standard therapy (MWA alone) as treatment for early stage HCC. Secondary aims are: 1) to determine the clinical feasibility of TAE + MWA in HCC patients with a small tumor burden using patient demographics and disease characteristic data and 2) to determine the effect of TAE on radiographic tumor characteristics in this patient cohort.

The primary outcome is 2-year intrahepatic disease-free survival, which is measured from time of randomization and is defined as the absence of local or regional recurrence of HCC as determined by diagnostic imaging. Local recurrence is defined as an enhancing lesion contiguous with the ablation zone that is present on subsequent imaging but was not present on the initial post-ablation scan. Regional recurrence is defined as hepatic recurrence that is not adjacent to the ablation site.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of hepatocellular carcinoma (HCC)
* HCC classification of stage 0 (very early) or stage A (early) according to Barcelona Clinic Liver Cancer (BCLC) staging system criteria
* Adequate clinical condition to undergo laparoscopic or robot-assisted laparoscopic transarterial embolization (TAE) and/or microwave ablation (MWA) as treatment for HCC
* Willing and able to give informed consent

Exclusion Criteria:

* Radiologic (computed tomography or magnetic resonance imaging) evidence of invasion into major portal/hepatic venous branches and no extrahepatic metastases
* Evidence of residual disease at first post-MWA computed tomography examination
* Body Mass Index (BMI) > 35
* Previous history of hepatic resections
* Severe renal dysfunction (creatinine clearance of <40 mL/min)
* Pregnant or nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dionisios Vrochides, MD PhD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Started | 5 | 3
Completed | 0 | 0
Not Completed | 5 | 3
Not completed — Physician Decision | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Median (Full Range); unit: years] | 62.4 [52 to 74] | 54.3 [51 to 59] | 59.4 [51 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 5 | 2 | 7
  Hispanic | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  American Indian/Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Asian | 0 | 0 | 0
  More Than One Race | 0 | 0 | 0
  Unknown / Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 3 | 8
BMI [Mean (Full Range); unit: kg/m^2] | 29.414 [25.9 to 33.7] | 28.57 [24.7 to 35.3] | 28.99 [24.7 to 35.3]
Consented Participants [Count of Participants; unit: Participants] | 5 | 3 | 8
Cirrhosis Present [Count of Participants; unit: Participants] | 5 | 3 | 8
Ascites Present [Count of Participants; unit: Participants] | 4 | 1 | 5
History of Hepatic Encephalopathy [Count of Participants; unit: Participants] | 3 | 0 | 3
History of Ascites [Count of Participants; unit: Participants] | 4 | 1 | 5
Please Note if any of the following are present (HCV, HPV, Heavy Alcohol use, drug use, nicotine use [Count of Participants; unit: Participants] | 4 | 3 | 7
Please Note if any previous treatment occured (colon: ablation, tace, chemo, embolization, resection [Count of Participants; unit: Participants] | 0 | 0 | 0
Please note any previous antiviral therapy the patient has received (IFN, PEG-IFN, Harvon, Other) [Count of Participants; unit: Participants] | 2 | 1 | 3
Method of diagnosis for HCC - CT [Count of Participants; unit: Participants] | 1 | 0 | 1
Method of diagnosis for HCC - MRI [Count of Participants; unit: Participants] | 4 | 3 | 7
Method of diagnosis for HCC - Biospy [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intrahepatic Disease-free Survival
Description: Defined as the absence of local or regional recurrence of hepatocellular carcinoma (HCC) as determined by diagnostic imaging
Time Frame: 2 years
Population: The analysis population description is not available. This study was terminated 1 year and 10 months after the enrollment of the first patient. There was not enough funding the support this study, and the PI opted to terminate the study.
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 5 | 3
Participants | 4 | 3

3. Secondary Outcome: Intrahepatic Disease-free Survival - 1 Year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 5 | 3
Participants | 4 | 3

4. Secondary Outcome: Postoperative Morbidity
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

5. Secondary Outcome: Postoperative Mortality
Time Frame: Assessed at 1 month and 3 months, total number up to 3 months reported
Measure: Count of Participants; unit: Participants
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

6. Secondary Outcome: Overall Survival
Time Frame: 2 Years
Population: as for outcome 1
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Survival - 3 Years
Time Frame: 3 Years
Population: as for outcome 1
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Survival - 5 Year
Time Frame: 5 Years
Population: as for outcome 1
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Intrahepatic Disease-free Survival - 2 Year
Description: Defined as the absence of local or regional recurrence of hepatocellular carcinoma (HCC) from date of treatment until 2 years after that date as determined by diagnostic imaging
Time Frame: 2 Year
Population: as for outcome 1
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Intrahepatic Disease-free Survival - 3 Year
Time Frame: 3 Year
Population: as for outcome 1
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Intrahepatic Disease-free Survival - 5 Year
Time Frame: 5 Year
Population: as for outcome 1
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Postoperative Morbidity
Time Frame: 3 Month
Measure: Count of Participants; unit: Participants
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
Number analyzed (Participants) | 5 | 3
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Arm/Group | TAE + MWA Combination Therapy | MWA Monotherapy
All-Cause Mortality (participants affected / at risk) | 2/5 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAE + MWA Combination Therapy (N=5) | MWA Monotherapy (N=3)
Hypotensive (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Difficulty with maintaining 02 stats and hypotensive after the MWA ablation on 8/12/2016, patient monitored in the ICU and later moved to the floor for observation.

LIMITATIONS AND CAVEATS:
Study closed early due to physician decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT02704130/Prot_SAP_000.pdf